CLINICAL TRIAL: NCT04493385
Title: Nationwide Hepatitis C NAT+ Cardiac Transplant Experience
Brief Title: The Hepatitis C Transplant Collaborative
Status: Recruiting | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 019-297
Record Dates: First submitted 2020-07-13; First posted 2020-07-30 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Transplant; Failure, Heart; Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study we seek to test the hypothesis that safety and clinical outcomes after cardiac transplantation utilizing HCV NAT+ donor organs as currently performed are acceptable.

DETAILED DESCRIPTION:
Organ offers from donors with prior or chronic hepatitis C virus (HCV) exposure have been historically underutilized for orthotopic heart transplantation because of the post-transplantation risks [1, 2]. The use of HCV antibody-positive (Ab+) donors was associated with attenuated survival benefit after heart transplant and increased coronary allograft vasculopathy in the era before new highly effective direct-acting antiviral agents (DAAs) were developed [3-5]. These DAAs target multiple steps in the HCV replication life cycle [6]. Newer, well-tolerated, oral direct-acting antivirals (DAAs) have recently been transforming thoracic transplant outcomes after donor-derived HCV transmission. Moreover, now that HCV nucleic-acid testing (NAT), a polymerase chain reaction (PCR)-based approach to detecting viral activity, is widely available and used on all US donor organs, transplant centers have more relevant information about the donor, allowing better risk assessments.

As a result, the utilization of HCV NAT+ donor hearts for transplantation is rapidly gaining momentum, with the obvious benefits of an enlarged donor pool [7]. Appropriately, clinical safety trials are currently underway, including a multicenter effort led by the PI of this proposal. Moreover, since the last ~2 years many transplant centers across the nation have started transplanting HCV NAT+ donor organs as standard of care. We estimate that the number of HCV+ cardiac transplants is quickly outpacing the number of trial participants. Hence, it is imperative that safety assessments and risk analyses 'catch up with the real world'.

ELIGIBILITY:
Inclusion Criteria:

1. Recipient of a proven HCV NAT+ donor heart.
2. Re-transplant patients will be included.

Exclusion Criteria:

1. Multi-organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cardiac transplant recipients utilizing HCV NAT+ donor organs
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-09-16 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Number of donor HCV nucleic-acid testing positive (HCV NAT+) cardiac transplantation | 6.5 years
  To assess the current status of donor HCV NAT+ cardiac transplantation via retrospective data collection.
Failure versus Cure Rate for HCV NAT+ Heart Transplants | 6.5 years
  sustained viral response (SVR)-12 (cure-rate) for HCV negative recipient
Rate of Primary graft dysfunction (PGD) | 30 days
  Rate of Expected Post-Transplant Risks
1 year mortality | 1 Year
  Number of deaths
Cellular graft rejection rate | 6.5 years
  Graft rejection rate
Antibody Mediated Rejection rate | 6.5 years
  Graft rejection rate

CONTACTS AND LOCATIONS:
Overall Officials: Shelley A Hall, MD FACC, Principal Investigator — BSWRI
Locations (1):
- Baylor Scott & White Health Research Institute, Dallas, Texas, United States

REFERENCES:
- [Background] Kim EY, Ko HH, Yoshida EM. A concise review of hepatitis C in heart and lung transplantation. Can J Gastroenterol. 2011 Aug;25(8):445-8. doi: 10.1155/2011/947838. PMID 21912770
- [Background] Englum BR, Ganapathi AM, Speicher PJ, Gulack BC, Snyder LD, Davis RD, Hartwig MG. Impact of donor and recipient hepatitis C status in lung transplantation. J Heart Lung Transplant. 2016 Feb;35(2):228-35. doi: 10.1016/j.healun.2015.10.012. Epub 2015 Oct 9. PMID 26615769
- [Background] Gasink LB, Blumberg EA, Localio AR, Desai SS, Israni AK, Lautenbach E. Hepatitis C virus seropositivity in organ donors and survival in heart transplant recipients. JAMA. 2006 Oct 18;296(15):1843-50. doi: 10.1001/jama.296.15.1843. PMID 17047214
- [Background] Haji SA, Starling RC, Avery RK, Mawhorter S, Tuzcu EM, Schoenhagen P, Cook DJ, Ratliff NB, McCarthy PM, Young JB, Yamani MH. Donor hepatitis-C seropositivity is an independent risk factor for the development of accelerated coronary vasculopathy and predicts outcome after cardiac transplantation. J Heart Lung Transplant. 2004 Mar;23(3):277-83. doi: 10.1016/S1053-2498(03)00148-7. PMID 15019636
- [Background] Lee R, Kottilil S, Wilson E. Sofosbuvir/velpatasvir: a pangenotypic drug to simplify HCV therapy. Hepatol Int. 2017 Mar;11(2):161-170. doi: 10.1007/s12072-016-9776-8. Epub 2016 Dec 7. PMID 27928718
- [Background] Asselah T, Boyer N, Saadoun D, Martinot-Peignoux M, Marcellin P. Direct-acting antivirals for the treatment of hepatitis C virus infection: optimizing current IFN-free treatment and future perspectives. Liver Int. 2016 Jan;36 Suppl 1:47-57. doi: 10.1111/liv.13027. PMID 26725897
- [Background] Gottlieb RL, Hall SA. The New Direct Antiviral Agents and Hepatitis C in Thoracic Transplantation: Impact on Donors and Recipients. Curr Transplant Rep. 2018;5(2):145-152. doi: 10.1007/s40472-018-0192-y. Epub 2018 Apr 10. PMID 29774177